CLINICAL TRIAL: NCT01449838
Title: Phase I Study of Colistin Methanesulfonate Sodium (CMS-Na) -A Randomized, Double Blind, Placebo Controlled, Single and Repeat Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of CMS-Na in Healthy Japanese Male Subjects -
Brief Title: Phase I Study of Colistin Methanesulfonate Sodium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114490
Record Dates: First submitted 2011-09-08; First posted 2011-10-10 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Infections, Pseudomonas
MeSH Terms: conditions — Pseudomonas Infections | interventions — colistinmethanesulfonic acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator): Subjects were administered single dose or twice daily for 2.5 days repeat dose of placebo by the intravenous route.
  Interventions: Drug: Saline
- Colistimethate sodium (Experimental): 2.5 milligrams (mg)/kilogram (kg) of CMS-NA (as colistin activity or 75,000 International Unit/kg) was administered as single dose or twice daily for 2.5 days repeat dose by the intravenous route.
  Interventions: Drug: Colistimethate sodium

INTERVENTIONS:
Drug: Colistimethate sodium — active
  Arms: Colistimethate sodium
Drug: Saline — placebo
  Arms: Saline

SUMMARY:
This is a clinical study protocol for a single centre, randomized, double blind, placebo controlled, single and repeat dose study to investigate the safety, tolerability and pharmacokinetics of intravenous dosing of Colistin Methanesulfonate Sodium (CMS-Na) in healthy Japanese male subjects.

Eighteen subjects will receive CMS-Na 2.5mg/kg (as colistin activity or 75,000 IU/kg) or placebo as a single dose and twice daily for 2.5 days by intravenous infusion.

Blood and urine samples for pharmacokinetics analysis will be taken at regular intervals after dosing. Safety will be assessed by measurement of vital signs, Echocardiogram (ECGs), safety laboratory data, renal function and review of adverse events.

ELIGIBILITY:
<Inclusion Criteria>

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
2. Japanese ethnic origin defined as having been born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese. Subjects should also have lived outside Japan for less than 10 years at the time of screening.
3. Male between 20 and 55 years of age inclusive, at the time of signing the informed consent.
4. Subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until completion of the follow-up visit.
5. Body weight 50 kg(inclusive) and BMI (body mass index)within the range 18.5 - 25 kg/m2 inclusive.
6. AST, ALT, alkaline phosphatase and bilirubin less than 1.5(inclusive)xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
7. Subjects with no clinically significant value of CLcr, NAG and beta-2 microglobulin judged by the investigator.
8. Average QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block taken from triplicate assessments at screening.
9. No clinically active and relevant abnormality on 12-lead ECG at screening.
10. Non-smokers (never smoked or not smoking for >6 months with <10 pack years history [Pack years = (cigarettes per day smoked/20) x number of years smoked])
11. A signed and dated written informed consent is obtained from the subject
12. The subject is capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form
13. Able to complete all study procedures and planned treatment periods. <Exclusion Criteria>

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates and benzodiazepines. The detection of drugs with a legitimate medical use would not necessarily be an exclusion to study participation.
2. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
3. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
4. A positive test for HIV antibody.
5. History of regular alcohol consumption within 3months of the study defined as:

   an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units. One unit is equivalent to a 285 mL glass of full strength beer or 425 mL schooner of light beer or 1 (30 mL) measure of spirits or 1 glass (100 mL) of wine (NHMRC Guidelines [NHMRC, 2001])
6. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
7. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
8. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
9. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
10. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
11. Unwillingness or inability to follow the procedures outlined in the protocol.
12. Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products prior to screening.
13. The subject has a known allergy or hypersensitivity to colistin or derived components.
14. Subject is kept under regulatory of judicial order in an institution.
15. Subject is mentally or legally incapacitated.
16. The subject's systolic blood pressure is outside the range of 90-140 mmHg or diastolic blood pressure is outside the range of 45-90 mmHg.
17. Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.

<Other Eligibility Criteria Considerations> To assess any potential impact on subject eligibility with regard to safety, the investigator must refer to the Prescribing Information (see Appendix 2, 3 and 4) for detailed information regarding warnings, precautions, contraindications, adverse events, and other significant data pertaining to the investigational product being used in this study.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-10-23 (Actual); Primary Completion 2010-12-09 (Actual); Study Completion 2010-12-09 (Actual)

PRIMARY OUTCOMES:
Profile of pharmacokinetics (PK) | Single dose and repeat dose day 3: pre-dose, 15min (m), 30m, 35m, 1,2,4,6,8,12,16,24,36 and 48h after the start of infusion. Repeat dose day 1 and day 2: pre-dose and 12h after the start of infusion.
  Maximum drug concentration (Cmax), Time of occurrence of Cmax (tmax), Terminal phase half-life(t1/2), Area under the concentration-time curve: AUC(0-inf), AUC(0-12), AUC(0-last), Clearance (CL), Fraction of urinary excretion (fe), Accumulation ratio (Ro and Rs).
Profile of safety (single) | Vital: -24h, pre-dose, 2,4,8,12,24,36,48h after the start of infusion. ECGs: -24h, pre-dose, 12, 24, 36 and 48h after the start of infusion. Clinical lab: pre-dose, 24 and 48h after the start of infusion. Adverse event: All study period.
  Vital signs, ECGs, clinical laboratory test and adverse events.
Profile of renal function | Single and repeat dose day 3: Pre-dose, 12, 24 36 and 48h after the start of infusion. Repeat dose day 1 and day 2:Pre-dose and 12h after the start of infusion. CLcr urine sampling: -24-0h of start of single dose and 24-36, 36-48h after d3 repeat dose
  Urinary β2-microglobulin, N-acetyl-β-D-glucosaminidase and creatinine clearance (CLcr).
Profile of safety (repeat day1 and 2) | Vital: pre-dose, 2,4,8,12 and14h after the start of infusion. ECGs: pre-dose and 12h after the start of infusion. Clinical lab: pre-dose. Adverse event: All study period.
  Vital signs, ECGs, clinical laboratory test and adverse events.
Profile of safety (repeat day 3) | Vital: pre-dose, 2,4,8,12,24,36,48h after the start of infusion. ECGs: pre-dose, 12, 24, 36 and 48h after the start of infusion. Clinical lab: pre-dose, 24 and 48h after the start of infusion. Adverse event: All study period.
  Vital signs, ECGs, clinical laboratory test and adverse events.

SECONDARY OUTCOMES:
Profile of urinary PK | Single dose and repeat dose day 3: 0-2, 2-4, 4-6, 6-12, 12-18, 18-24, 24-30, 30-36, 36-42, 42-48h. Repeat dose day 1 and day 2: Every 6 hours.
  Urinary recovery (Ae) and Renal clearance (CLr)
Profile of other PK | Single dose and repeat dose day 3: pre-dose, 15m, 30m, 35m, 1,2,4,6,8,12,16,24,36 and 48h after the start of infusion. Repeat dose day 1 and day 2: pre-dose and 12h after the start of infusion.
  AUC(0-24), %AUCex, rambda_z, Volume of destribution based on the terminal phase (Vz) and volume of distribution at steady state (Vss)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

REFERENCES:
- [Result] Mizuyachi K, Hara K, Wakamatsu A, Nohda S, Hirama T. Safety and pharmacokinetic evaluation of intravenous colistin methanesulfonate sodium in Japanese healthy male subjects. Curr Med Res Opin. 2011 Dec;27(12):2261-70. doi: 10.1185/03007995.2011.626557. Epub 2011 Oct 14. PMID 21995648
- See also: Results for study 114490 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114490?search=study&search_terms=114490#rs